CLINICAL TRIAL: NCT02570022
Title: Liposomal Bupivacaine Versus Interscalene Nerve Block for Pain Control After Shoulder Arthroplasty: A Prospective Randomized Trial
Brief Title: Liposomal Bupivacaine in Total Shoulder Arthroplasty
Acronym: EXP-TSA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Kelechi Okoroha, Sub-Investigator, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LB-TSA
Record Dates: First submitted 2015-10-05; First posted 2015-10-07 (Estimated); Results first posted 2016-10-13 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-08

CONDITIONS: Pain
Keywords: Pain control; liposomal bupivacaine; exparel; shoulder arthroplasty
MeSH Terms: conditions — Pain; Agnosia | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liposomal bupivacaine (Experimental): Patients in this group received local infiltration of Liposomal bupivacaine before the end of surgery.
  Interventions: Drug: Liposomal bupivacaine
- Inter-scalene nerve block (Active Comparator): Patients in this group received preoperative ultrasound guided inter-scalene nerve blocks by senior anesthesiologist using ropivicaine.
  Interventions: Procedure: Inter-scalene nerve block; Drug: Ropivacaine

INTERVENTIONS:
Drug: Liposomal bupivacaine — Local infiltration of liposomal bupivacaine
  Other Names: exparel
  Arms: Liposomal bupivacaine
Procedure: Inter-scalene nerve block — Pre-operative inter-scalene nerve block
  Other Names: Naropin
  Arms: Inter-scalene nerve block
Drug: Ropivacaine — Ropivicaine was used for the inter-scalene nerve block.
  Arms: Inter-scalene nerve block

SUMMARY:
This is a randomized, single blinded, standard of care controlled clinical trial. All adult patients over eighteen desiring shoulder arthroplasty will be eligible. The study compares pain control and opioid consumption in patients undergoing shoulder arthroplasty between patients receiving liposomal bupivacaine and those who underwent a preoperative inter-scalene nerve block.

DETAILED DESCRIPTION:
Study Design: A randomized single blinded standard of care controlled clinical trial comparing pain management interventions. All patients over age eighteen and scheduled for primary shoulder arthroplasty (SA) a three fellowship trained surgeons will be eligible for inclusion. Patients will be excluded if their medical history presents known allergies or intolerance to dexamethasone, opioid or bupivacaine, substantial alcohol or drug abuse, and pregnancy.

Liposomal Bupivacaine has a refrigerated shelf life of one month the investigational facility. Patients will be sequentially recruited into the randomization process. Liposomal Bupivacaine will be held by the Henry Ford hospital pharmacy up to one month prior to planned shoulder arthroplasty in anticipation of surgery on eligible patients. The sterile solutions will be delivered to and kept by the inpatient clinical pharmacy until the date of surgery and delivered to the operating room at the beginning of a surgical case. The current dose of Liposomal Bupivacaine has been chosen based on previously published data of local infiltrative analgesia with Liposomal Bupivacaine and one published study on Liposomal Bupivacaine efficacy.

The week prior to surgery, patients will be randomized to receive Local infiltration anesthesia (LIA) with Liposomal Bupivacaine, or Inter-scalene nerve block (INB) using a computer generated sequence. The results of randomization will be securely delivered to the anesthesiologist and the surgeon the week prior. The anesthesiologist will view the assigned group to determine if a preoperative INB will be given. Depending on the randomization group either an Liposomal Bupivacaine solution will be delivered to the operating room for local infiltration or the anesthesiologist will perform a preoperative INB.

Patients in the Liposomal Bupivacaine group will receive LIA with 10cc(133mg) of Liposomal Bupivacaine solution dissolved in 20cc of sterile saline before wound closure. The solution will be applied to the wound bed, muscles, and periosteum. The solution will be left unperturbed for five minutes. Thereafter the solution will be suctioned from the wound and the shoulder joint. Incisions will be closed in typical fashion and the wound dressed.The tourniquet will be deflated.

Patients in the INB will receive postoperative ultrasound guided INB. Experienced anesthesiologists will apply all INBs in this study.

Following the procedure pain will be accessed subjectively through visual analog scale and numeric rating scale pain scores, pain diaries given to the patient to record at home, pain summary scores at follow up visits and objectively through narcotic pain requirement. A blind observer will also access outcomes.

Planned Data Analysis:

Means and standard deviations, as well as medians and interquartile ranges will be computed for pain scores.These outcomes will be compared by Wilcoxon rank sum tests. The amount of pain medication and pain scores will be compared by Wilcoxon rank sum tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 scheduled for primary shoulder arthroplasty by three fellowship trained surgeons will be eligible for inclusion

Exclusion Criteria:

* Patients will be excluded if their medical history presents known allergies or intolerance to dexamethasone, opioid or bupivacaine, substantial alcohol or drug abuse, and pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-10; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liposomal Bupivacaine | Inter-scalene Nerve Block
Started | 26 | 31
Completed | 26 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Sixty patients were recruited for the study. Three patients declined to participate and were excluded before randomization. The remaining 57 patients were randomized with 31 patients in the INB group and 26 patients in the LB group. No patients were lost to follow-up. There were no statistical differences in any demographics between the 2 groups
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivacaine | Inter-scalene Nerve Block | Total
Number analyzed (Participants) | 26 | 31 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 27 | 47
  >=65 years | 6 | 4 | 10
Age, Continuous [Mean (Full Range); unit: years] | 69.4 [50 to 75] | 67.1 [49 to 86] | 67.8 [49 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 12 | 16 | 28
Region of Enrollment [Number; unit: participants]
  United States | 26 | 31 | 57

OUTCOME MEASURES:

1. Primary Outcome: Pain Levels
Description: Patients recorded pain levels every four hours using Visual analog scales for four days post operatively. Average daily pain was calculated for each patient. Range of the visual analog scale was 0-10, where 0 indicated a lower amount of pain and 10 indicated higher amount of pain.
Time Frame: four days postoperatively
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Liposomal Bupivacaine | Inter-scalene Nerve Block
Number analyzed (Participants) | 26 | 31
units on a scale
  Mean Pain score Day 0 | 4.8 (1.8) | 4.0 (1.8)
  Mean Pain score Day 1 | 4.7 (2.3) | 4.0 (1.7)
  Mean Pain score Day 2 | 4.3 (2.5) | 3.6 (1.7)
  Mean Pain score Day 3 | 4.1 (2.0) | 4.3 (2.1)
Statistical Analysis 1: Comparison: Liposomal Bupivacaine vs Inter-scalene Nerve Block; Our hypothesis was that in patients undergoing shoulder arthroplasty, treatment with LB would lead to no significant differences in average daily pain scores. A power analysis was performed prior to the study to assess the primary hypothesis that a significant difference in average daily pain of 13mm on VAS will not be found between the INB and LB groups. With a power of 80% (beta level = 0.80, alpha level = 0.05), a sample size of 25 patients per group was obtained; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.05 — This analysis corresponds to the visual analog scale and morphine equivalent data

2. Secondary Outcome: Morphine Equivalents
Description: Patients recorded opioid intake for four days postoperatively. Patients average daily morphine consumption was determined by averaging total patients daily morphine consumption by the number of patients.
Time Frame: four days postoperatively
Measure: Mean (Standard Deviation); unit: mg of morphine equivalent
Arm/Group | Liposomal Bupivacaine | Inter-scalene Nerve Block
Number analyzed (Participants) | 26 | 31
mg of morphine equivalent
  Mean Morphine equivalents used Day 0 | 14.8 (9.2) | 21.4 (11.3)
  Mean Morphine equivalents used Day 1 | 8.9 (9.7) | 9.1 (11.4)
  Mean Morphine equivalents used Day 2 | 12.3 (16.9) | 5.2 (10.8)
  Mean Morphine equivalents used Day 3 | 2.8 (4.1) | 2.2 (6.1)

ADVERSE EVENTS:
Arm/Group | Liposomal Bupivacaine | Inter-scalene Nerve Block
Serious Adverse Events (participants affected / at risk) | 0/26 | 1/31
Other Adverse Events (participants affected / at risk) | 0/26 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liposomal Bupivacaine (N=26) | Inter-scalene Nerve Block (N=31)
Phrenic nerve palsy (Nervous system disorders) | 0 (0) | 1 (1) — One patient in the INB group suffered a prolonged phrenic nerve palsy requiring readmission for elevation of the right hemi-diaphragm with respiratory compromise.

LIMITATIONS AND CAVEATS:
Use of the VAS, which is a simple one-dimensional analog rating scale, to assess the patients subjective pain level. Patient compliance is a limitation, with maintenance of pain dairies decreasing as time from surgery progressed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No